CLINICAL TRIAL: NCT04113122
Title: Senescence and the Early Ageing Phenotype After Chemotherapy for Testicular Cancer: the SEA-CAT Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 201700615
Record Dates: First submitted 2019-01-08; First posted 2019-10-02 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Intervention Model Description: A study will be performed consisting of two cohorts. Cross-sectional study Testicular cancer survivors treated between 2000 and 2005 or between 2006 and 2012 with cisplatin-combination chemotherapy and were extensively phenotypically mapped within two longitudinal trials will be invited to participate in a single cross-sectional follow-up study visit 5-20 years after chemotherapy.
  Longitudinal study
  Patients with metastasized testicular cancer who are about to start with cisplatin-combination chemotherapy will be invited. Study participation involves four study visits:
  Visit 1: before start of chemotherapy Visit 2: before third cycle of chemotherapy Visit 3: one month after completion of chemotherapy Visit 4: one year after start of chemotherapy
  Patients with stage I testicular cancer will serve as control group with three study visits:
  Visit 1: at time of orchidectomy Visit 2: one month after orchidectomy Visit 3: one year after orchidectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cross-sectional study: (Experimental): Testicular cancer survivors who were treated between 2000 and 2005 or between 2006 and 2012 with cisplatin-combination chemotherapy and who were extensively phenotypically mapped within two longitudinal trials (15,16) will be invited to participate in a single cross-sectional follow-up study visit 5-20 years after chemotherapy.
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Subcutaneous fat biopsy
- Longitudinal study - chemotherapy group (Experimental): Patients with metastasized testicular cancer who are about to start with cisplatin-combination chemotherapy will be invited in the longitudinal part of this study. Study participation involves four study visits:
  Visit 1: before start of chemotherapy Visit 2:before third cycle of chemotherapy Visit 3: one month after completion of chemotherapy Visit 4: one year after start of chemotherapy
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Subcutaneous fat biopsy
- Longitudinal study - stage I control group (Other): Patients with stage I testicular cancer will serve as control group with three study visits:
  Visit 1: at time of orchidectomy Visit 2: one month Visit 3: one year after orchidectomy
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Subcutaneous fat biopsy

INTERVENTIONS:
Diagnostic Test: Skin biopsy — A 4 mm skin biopsy will be performed at the upper leg of the patient. Before the skin biopsy local anesthesia is applied subcutaneously. In these skin biopsies senescent cells will be detected by p16, p21 and yH2Ax staining. Furthermore, we will measure platinum levels in the skin biopsies.
Diagnostic Test: Subcutaneous fat biopsy — An abdominal subcutaneous fat biopsy will be performed 7-10 cm on the right side of the umbilicus. Before the fat biopsy local anesthesia is applied subcutaneously. An amount of 30 mg fat tissue will be collected using needle aspiration.
  In these fat biopsies senescent cells will be detected by p16, p21 and yH2Ax staining. Furthermore, we will measure platinum levels (ICP-MS), adipocytokines (leptin, adiponectin, interleukin-6, PAI-1, TNF-α), p53 activation indirectly by measuring p21 or mdm2 expression using immunohistochemistry, microRNA regulation of insulin signaling in adipose tissue: miR-103, miR-107, miR-29.

SUMMARY:
Cisplatin-combination chemotherapy causes inevitably DNA damage by platinum-DNA adduct formation of both tumor cells but also healthy cells. It therefore stands to reason that testicular cancer treatment causes an increased burden of senescent cells, which causes upregulation of the SASP resulting in a pro-inflammatory phenotype. The investigators hypothesize that this may be an important mechanism behind development of late effects and an early ageing phenotype after treatment for testicular cancer.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the cross-sectional part of this study, a subject must meet all of the following criteria:

* Diagnosed with metastatic testicular cancer in 1999-2012 (stage II or higher)
* Received first-line cisplatin-based chemotherapy
* Was younger than 50 years of age at start of chemotherapy

In order to be eligible to participate in the longitudinal part of this study, a subject must meet all of the following criteria:

Chemotherapy-group:

* Diagnosis of metastatic testicular cancer (stage II or higher)
* Is about to start with first-line cisplatin-based chemotherapy
* Younger than 50 years of age at diagnosis of metastatic testicular cancer

Stage I control-group:

* Diagnosis of testicular cancer stage I disease
* Younger than 50 years of age at diagnosis of testicular cancer

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

- Not able to provide informed consent (in example in case of mental or psychiatric disability)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-02-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cellular senescence | 1 year
  The change in the amount of senescent cells in skin and fat tissue (defined as % of cells in which nucleus is stained positive for P16, P21 and yH2Ax)

SECONDARY OUTCOMES:
Senescence-associated secretory phenotype (SASP) | 1 year
  Change in levels of the cytokines: IL-6, IL-8, VEGF
Pulse-wave velocity | 1 year
  Presence or development of the early ageing phenotype will be assessed measuring vascular damage: change in vascular stiffness (pulse-wave velocity, PWV).
Platinum levels | 1 year
  Changes in circulating platinum levels and the amount of platinum depositions in skin and fat tissure will be assessed.
Adipocytokines 1 | 1 year
  Changes in levels of leptin and PAI-1 (ug/L)
Adipocytokines 2 | 1 year
  Changes in levels of adiponectin (ug/mL)

CONTACTS AND LOCATIONS:
Overall Officials: J. A. Gietema, Prof., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands